CLINICAL TRIAL: NCT06686875
Title: Assessment of the Prevalence of Persistent Postoperative Pain in Patients Undergoing Laparoscopic Gastrectomy
Brief Title: Chronic Abdominal Pain After Laparoscopic Sleeve Gastrectomy
Acronym: Chron Pain LSG
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Mieszczanski, Principal Investigator, Medical University of Warsaw
Other Study IDs: AKBE/266/2024
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Chronic Pain; Abdominal Pain
Keywords: laparoscopic sleeve gastrectomy; chronic postoperative pain; neuropathic pain
MeSH Terms: conditions — Obesity; Chronic Pain; Abdominal Pain; Pain, Postoperative; Neuralgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Post surgical group
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients will receive a link to a web-based questionnaire on the prevalence and characteristics of pain symptoms including the PainDETECT questionnaire.

SUMMARY:
The study aims to evaluate the prevalence of postoperative chronic pain, defined as the persistence of abdominal pain for more than 3 months after laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
The main goal of this study is to determine the incidence of chronic abdominal pain among patients who have undergone laparoscopic sleeve gastrectomy. Patients who underwent this type of surgery at the Department of General Surgery and Transplantology of the Medical University of Warsaw between January 2020 and August 2024 will be qualified for the study. The participants will be asked to complete an online questionnaire, including a pain scale and PainDETECT Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent laparoscopic sleeve gastrectomy 3 months to 5 years earlier

Exclusion Criteria:

* Lack of patient consent to participate in the survey
* No possibility to contact the patient
* Revisional procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent surgery at the Department of General Surgery and Transplantology of the Medical University of Warsaw between January 2020 and December 2024
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
The presence of chronic abdominal pain after laparoscopic sleeve gastrectomy | Baseline
  The presence of pain after laparoscopic sleeve gastrectomy, which persists more than 3 months postoperatively.

SECONDARY OUTCOMES:
PainDETECT Questionnaire score | Baseline
  PainDETECT is a simple, easy-to-use screening questionnaire. The questionnaire consists of 9 items and is completed by the patient. There are 7 weighted sensory descriptor items (never to very strongly) and 2 items relating to spatial and temporal pain characteristics. A total score of 19 or more is indicative of likely neuropathic pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University in Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mieszczanski P, Jurczak M, Kolacz M, Gorniewski G, Godlewska I, Ziemianski P, Cylke R, Lisik W, Trzebicki J. Chronic Post-Surgical Pain After Laparoscopic Sleeve Gastrectomy: Is the Opioid-Free Anesthesia Superior? A Cross-Sectional Study. J Clin Med. 2025 Oct 30;14(21):7721. doi: 10.3390/jcm14217721. PMID 41227115